CLINICAL TRIAL: NCT02003352
Title: Evaluation of the Effectiveness of a Novel Brain and Vestibular Rehabilitation Treatment Modality in PTSD Patients Who Have Suffered Combat Related Traumatic Brain Injuries
Brief Title: Study of PTSD in Military Veterans Who Have Suffered Traumatic Brain Injuries
Acronym: PTSD-TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carrick Institute for Graduate Studies (Other)
Collaborators: Carrick Brain Centers (Industry)
Responsible Party: Principal Investigator, Frederick Carrick, PhD, FACCN, Principal Investigator, Carrick Institute for Graduate Studies
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBC11013
Record Dates: First submitted 2013-10-29; First posted 2013-12-06 (Estimated); Results first posted 2017-03-23 (Actual); Last update posted 2017-03-23 (Actual); Status verified 2017-01

CONDITIONS: PTSD; TBI
Keywords: TBI; PTSD; Functional Neurology; Vestibular Rehabilitation; Dynamic Computerized Posturography; Saccadometry
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Functional Neurological Rehabilitation (Experimental): Functional Neurological and physical/vestibular rehabilitation strategies
  Interventions: Procedure: Functional Neurological Rehabilitation

INTERVENTIONS:
Procedure: Functional Neurological Rehabilitation — Functional Neurological Rehabilitation Includes vestibular rehabilitation and physical rehabilitation. Vestibular rehabilitation utilizes strategies that involves movement of the head and eyes at various speeds and directions while the subject looks at a target. Physical rehabilitation involves exercises to increase mobility and increase strength.

SUMMARY:
Treatment for veterans who have had a traumatic brain injury (TBI) and who are suffering from post traumatic stress syndrome (PTSD) is varied with varied outcomes. Investigators will study PTSD treatment in military Veterans who have suffered traumatic brain injuries. Investigators will use 1 independent specialty treatment centers that utilize a specific novel methodology of PTSD treatments and study the clinical outcomes of veterans who have suffered a TBI with associated post-concussive symptoms and other comorbidities such as PTSD. Investigators hypothesize that the treatment of PTSD will have a significant outcome with neurological physical and vestibular rehabilitation when compared to psychological or psychiatric therapy. This study will use gold standard measurement scales and compare changes in the scales after treatment to evaluate the treatments.

DETAILED DESCRIPTION:
The Department of Defense and the Defense and Veteran's Brain Injury Center estimate that 22% of all combat casualties from conflicts in Iraq and Afghanistan are brain injuries. Patients with TBI often meet criteria for PTSD on screening instruments for TBI and vice versa. No screening instruments available can reliably make the diagnosis of PTSD and the gold standard remains an interview by a skilled clinician using the Clinician-Administered PTSD Scale (CAPS) a 30-item structured interview that corresponds to the Diagnostic and Statistical Manual of Mental Disorders IV (DSM-IV) criteria for PTSD. Treatment for veterans who have had a TBI and who are suffering from PTSD is varied with varied outcomes. Investigators propose a Randomized Prospective Clinical Trial of PTSD treatment in military Veterans that have suffered traumatic brain injuries. Investigators will use 2 independent specialty treatment centers that utilize different methodology of PTSD treatments and study the clinical outcomes of veterans who have suffered a TBI with associated post-concussive symptoms and other comorbidities such as PTSD. This study will use a baseline CAPS assessment and investigators will establish cut points and randomize from within those to establish a stratified randomization within groups. Subjects will undergo treatments and an outcome CAPS score will be obtained at the end of treatment as the primary outcome to calculate if there is a change in score that is statistically or clinically significant. Investigators also will utilize secondary outcomes to measure any changes in the scores obtained by these instruments. These instruments and measures such as Computerized Dynamic Posturography and video electronystagmography and saccadometry will be obtained before the initiation of treatment and when treatment is terminated to measure a change in score. All instruments will be used to measure changes in function that are related to changes in PTSD symptomatology and neurological function

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PTSD
* History of Traumatic Brain Injury
* Military veteran of conflict in war zone

Exclusion Criteria:

* Criminal history of violence

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2014-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick R Carrick, PhD, Principal Investigator — Carrick IGS
Locations (1):
- Carrick Brain Centers, Irving, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carrick FR, McLellan K, Brock JB, Randall C, Oggero E. Evaluation of the Effectiveness of a Novel Brain and Vestibular Rehabilitation Treatment Modality in PTSD Patients Who have Suffered Combat-Related Traumatic Brain Injuries. Front Public Health. 2015 Feb 4;3:15. doi: 10.3389/fpubh.2015.00015. eCollection 2015. PMID 25699246
- [Derived] Carrick FR, Pagnacco G, McLellan K, Solis R, Shores J, Fredieu A, Brock JB, Randall C, Wright C, Oggero E. Short- and Long-Term Effectiveness of a Subject's Specific Novel Brain and Vestibular Rehabilitation Treatment Modality in Combat Veterans Suffering from PTSD. Front Public Health. 2015 Jun 1;3:151. doi: 10.3389/fpubh.2015.00151. eCollection 2015. PMID 26082920

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Functional Neurological Rehabilitation
Started | 98
Completed | 98
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Functional Neurological Rehabilitation: Functional Neurological and physical/vestibular rehabilitation strategies
  Functional Neurological Rehabilitation: Functional Neurological Rehabilitation Includes vestibular rehabilitation and physical rehabilitation. Vestibular rehabilitation utilizes strategies that involves movement of the head and eyes at various speeds and directions while the subject looks at a target. Physical rehabilitation involves exercises to increase mobility and increase strength.
  The study population consisted of 98 combat veterans who had suffered aT BI with PTSD, referred to our study by Veteran's groups. All subjects were male with a mean age of 39 years with a minimum age of 20 years and a maximum age of 60 years.They all met the inclusion requirements and did not have any of the exclusion requirements.
Arm/Group | Functional Neurological Rehabilitation
Number analyzed (Participants) | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 98
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 39 [20 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 98
Region of Enrollment [Number; unit: participants]
  United States | 98

OUTCOME MEASURES:

1. Primary Outcome: Change in Diagnostic and Statistical Manual of Mental Disorders IV Clinician-Administered PTSD Scale DSM IV-(CAPS)
Description: The CAPS is the gold standard in PTSD assessment and is a 30-item structured interview.For each symptom, standardized questions and probes are provided. Administration requires identification of an index traumatic event to serve as the basis for symptom inquiry. The full interview takes 45-60 minutes to administer.CAPS symptom severity ratings are based on symptom frequency and intensity (except for amnesia and diminished interest which are based on amount and intensity). Higher scores represent a worse outcome with severity categories of 0-19 (minimal), 20-39 (mild), 40-59 (moderate), 60-79 (severe), 80-136 (extreme). We will use changes in the DSM-IV CAPS scores before and after treatment to distinguish between the estimated frequency and intensity of the various symptoms. Frequency and intensity scores will be combined to give a total CAPS score (range: 0-136) CAPS testing was scheduled pre-intervention, 1 week post-intervention, and at 3 months post-intervention.
Time Frame: up to 12 weeks
Population: Changes in CAPS scores before-after. Frequency and intensity scores combined-CAPS score (range: 0-136) . CAPS pre-intervention, 1 week post-intervention, and at 3 months post-intervention. Difference pre and post of CAPS Scores (matched pairs) two-tailed t -Test with alpha of <0.05. Effect Size Cohen's D
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Functional Neurological Rehabilitation
Number analyzed (Participants) | 98
units on a scale | 73.13 [69.17 to 77.09]

ADVERSE EVENTS:
Arm/Group | Functional Neurological Rehabilitation
Serious Adverse Events (participants affected / at risk) | 0/98
Other Adverse Events (participants affected / at risk) | 0/98

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes